CLINICAL TRIAL: NCT04630054
Title: Can Face Masks Reduce Transmission of SARS-CoV-2 in Bangladesh? A Cluster Randomized Controlled Trial
Brief Title: Face Masks to Reduce COVID-19 in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Stanford University (Other); Innovations for Poverty Action (Other); North South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000028482
Record Dates: First submitted 2020-11-13; First posted 2020-11-16 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Covid19
Keywords: Masks; Transmission; Seroprevalence; Bangladesh
MeSH Terms: conditions — COVID-19 | interventions — Masks

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The intervention involves wearing a face mask so participants will know if they are in the intervention group. The investigators will be blinded as to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mask Intervention (Experimental): Communities and individuals randomized to the intervention arm will be given masks and behavior change communication to motivate proper mask use.
  In the community experiment, every adult in communities randomized to the intervention arm will be encouraged to wear a mask when outside their housing compound and around other people.
  In the individual experiment, individuals randomized to the intervention arm will not be asked to recommend masks to others, but will also not be discouraged from recommending mask use to others.
  Interventions: Device: Face mask; Behavioral: Face mask awareness
- Control (No Intervention): Control individuals will receive no masks or behavior change communication.

INTERVENTIONS:
Device: Face mask — Intervention individuals will be given cloth or surgical face masks.
  Arms: Mask Intervention
Behavioral: Face mask awareness — Intervention individuals will be told about the importance of wearing face masks that cover the nose, mouth, and chin. Mask by mask promoters and community and religious leaders will encourage mask wearing.
  Arms: Mask Intervention

SUMMARY:
The primary goal of the village-level intervention is to assess whether mask-wearing reduces community-level COVID-19 seroconversion. The individual experiment assess whether masks protect against COVID-19 seroconversion. It also assesses the efficacy of high-quality cloth vs. surgical masks.

DETAILED DESCRIPTION:
This study intends to answer the following research questions:

Can mask distribution and mask promotion at homes, mosques, markets and other public areas successfully change community mask-wearing norms to increase mask-wearing?

Can community mask-wearing reduce COVID-19 seroconversions?

Can mask wearing reduce COVID-19 seroconversions for the wearer?

Are high-quality cloth or "surgical" masks more effective in reducing COVID-19 seroconversions?

Is increased prevalence of community-level mask-wearing associated with decreased physical distancing?

To answer these questions, the investigators will conduct a cluster randomized trial which randomizes the proposed intervention at the village level in Bangladesh, as well as a separate trial where masks are randomized at the individual level among high-risk indoor market vendors.

In the community experiment, control communities will receive no intervention and treatment communities will receive an extensive intervention combining several elements. The investigators will distribute free face masks through door-to-door visits and at markets and mosques. Some communities will receive cloth masks and some will wear surgical masks (cross-randomized among intervention communities). Mask promoters in the community and at markets in treated villages will remind people about the importance of wearing masks and distribute additional masks. Markets will have signs that masks need to be worn to enter the market. Religious leaders will encourage mask use at religious services. Communities will receive an incentive if >75% are observed to wear masks by mask surveillance staff that conduct discrete observations on days when mask promotion is and is not occurring. The project will enroll 600 communities and create matched pairs based on population size; half of which will be randomized to receive the intervention.

In the individual experiment, the investigators will identify 5,000 high-risk individuals (vendors at indoor market). and randomizing them at the individual level to receive our mask intervention or not. In each indoor market, there will be both control and treatment individuals. Individuals in the treatment arm will receive a free face mask (cloth or surgical). Investigators will enroll individuals from 350-500 markets that are not in the communities that are participating in the community experiment.

Communities will be surveilled at 0, 1, 2, 4, 6, 8, and 12 weeks to assess mask wearing. Participants in the indvidual experiment will be surveilled at 0, 1, 2, 4, 6, weeks to assess mask wearing.

In both experiments, we will assess seroprevalence of COVID-19 at baseline and endline. Endline is planned for 12 weeks after the intervention begins, but may be shifted according to seroprevalence trends.

ELIGIBILITY:
Inclusion Criteria:

* Community experiment: Live in selected village
* Individual experiment: Work in selected market

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350000 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Symptomatic SARS-CoV2 infection | 12 weeks
  Symptomatic SARS-CoV2 infection, assessed via antibody testing 12 weeks after baseline, among individuals who report symptoms consistent with COVID-19 at 5 weeks or 9 weeks after baseline

SECONDARY OUTCOMES:
SARS-CoV2 infection | 12 weeks
  Community experiment: Symptomatic SARS-CoV2 infection, assessed via antibody testing 12 weeks after baseline relative to baseline tests, among 25,000 high-risk individuals from randomly selected households
  Individual experiment: Symptomatic SARS-CoV2 infection, assessed via serological testing 10 weeks after baseline, among all 5,000 individuals in individual experiment
Observed prevalence of proper mask wearing | intervention weeks 0, 1, 2, 4, 6, 8, and 12 in the community experiment and intervention weeks 0, 1, 2, 4, and 6 in the individual experiment
  Wearing a mask of the nose, mouth, and chin
Respiratory infection prevalence | 5 and 9 weeks
  Prevalence of self-reported symptoms of COVID-19, including fever, cough, sore throat, shortness of breath, difficulty breathing, nasal congestion, and runny nose.

CONTACTS AND LOCATIONS:
Locations (1):
- Innovations for Poverty Action, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data with other researchers

REFERENCES:
- [Derived] Constantin AM, Noertjojo K, Sommer I, Pizarro AB, Persad E, Durao S, Nussbaumer-Streit B, McElvenny DM, Rhodes S, Martin C, Sampson O, Jorgensen KJ, Bruschettini M. Workplace interventions to reduce the risk of SARS-CoV-2 infection outside of healthcare settings. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD015112. doi: 10.1002/14651858.CD015112.pub3. PMID 38597249
- [Derived] Abaluck J, Kwong LH, Styczynski A, Haque A, Kabir MA, Bates-Jefferys E, Crawford E, Benjamin-Chung J, Raihan S, Rahman S, Benhachmi S, Bintee NZ, Winch PJ, Hossain M, Reza HM, Jaber AA, Momen SG, Rahman A, Banti FL, Huq TS, Luby SP, Mobarak AM. Impact of community masking on COVID-19: A cluster-randomized trial in Bangladesh. Science. 2022 Jan 14;375(6577):eabi9069. doi: 10.1126/science.abi9069. Epub 2022 Jan 14. PMID 34855513

DOCUMENTS (3):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT04630054/Prot_004.pdf
  • Statistical Analysis Plan (2021-06-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT04630054/SAP_002.pdf
  • Informed Consent Form (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT04630054/ICF_003.pdf